CLINICAL TRIAL: NCT03752437
Title: Comparison of Two Dosages of Heparin Before Extracorporeal Circulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Head of Department, Astes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MDKR
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Extracorporeal Circulation; Complications
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Intervention Model Description: One arm will receive 300 IU of heparin based on real weight, and the other arm will receive 300 IU of heparin based on ideal weight.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomisation by computer, different sheet for encoding data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Weight (Experimental): Injection of 300 IU of heparin based on REAL weight. This injection will be controlled by an ACT (activated clotting time) one minute after the injection.
  Interventions: Diagnostic Test: ACT (Activated Clotting Time); Drug: Heparin
- Ideal Weight (Experimental): Injection of 300 IU of heparin based on IDEAL weight. This injection will be controlled by an ACT (activated clotting time) one minute after the injection.
  Interventions: Diagnostic Test: ACT (Activated Clotting Time); Drug: Heparin

INTERVENTIONS:
Diagnostic Test: ACT (Activated Clotting Time) — Measure of ACT in the two arms in order to determine if injection of heparin based on ideal weight is better or not than those one on real weight.
Drug: Heparin — 300 IU of heparin

SUMMARY:
In this study the investigators will study two dosages of heparin before extracorporeal circulation in open chest cardiac surgery.

DETAILED DESCRIPTION:
In this study the investigators will study two dosages of heparin before extracorporeal circulation in open chest cardiac surgery. The first dosage will be 300 IU per kilogram of REAL weight, the second dosage will be 300 IU per kilogram of IDEAL weight.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for cardiac open chest surgery

Exclusion Criteria:

* Patient's refusal
* Antithrombin III factor < 75%
* Patient under treatment by heparin IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
ACT performance | 1 minute
  Measure of ACT to be > 400 seconds to allow extracorporeal circulation, but also < 700 seconds to avoid excessive bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, PhD, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc of Bouge, Namur, Belgium